CLINICAL TRIAL: NCT03482648
Title: A Phase I, Randomized, Double-Blind, Placebo-Controlled Study to Evaluate Safety, Tolerability and Pharmacokinetics of Novel Oral Peptide BBT-401-1S Following Single and Multiple Ascending Doses in Healthy Adult Subjects
Brief Title: First-In-Human Study of BBT-401-1S Following Single and Multiple Ascending Doses in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bridge Biotherapeutics, Inc. (Industry)
Collaborators: KCRN Research, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BBT401-UC-US01
Record Dates: First submitted 2018-03-17; First posted 2018-03-29 (Actual); Last update posted 2021-07-21 (Actual); Status verified 2021-07

CONDITIONS: Ulcerative Colitis
Keywords: Pellino-1
MeSH Terms: conditions — Colitis, Ulcerative

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Single Ascending Doses (Experimental)
  Interventions: Drug: BBT-401-1S, Single dose; Drug: Placebo
- Multiple Ascending Doses (Experimental)
  Interventions: Drug: BBT-401-1S, Multiple doses; Drug: Placebo

INTERVENTIONS:
Drug: BBT-401-1S, Single dose — Single dose of BBT-401-1S, 7 dose levels, oral capsule
  Arms: Single Ascending Doses
Drug: BBT-401-1S, Multiple doses — Multiple doses of BBT-401-1S, 7 days, 3 dose levels, oral capsule
  Arms: Multiple Ascending Doses
Drug: Placebo — Placebo matched to BBT-401-1S, oral capsule

SUMMARY:
This clinical trial is the first-in-human study of BBT-401-1S. The purpose of this phase 1 study is to assess the safety and tolerability of single and multiple ascending oral doses of BBT-401-1S in healthy adult subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy adult male and/or female (non-childbearing potential only), 19 to 55 years of age, inclusive, at screening.
2. Continuous non-smoker who has not used nicotine-containing products for at least 3 months prior to the first dose and throughout the study.
3. Body mass index (BMI) ≥ 18.5 and ≤ 32.0 (kg/m2) at screening and weight ≥ 50 kg at screening.
4. Medically healthy with no clinically significant medical history, physical examination, laboratory profiles, vital signs or ECGs, as deemed by the PI.
5. No clinically significant history or presence of ECG findings as judged by the PI or qualified designee at screening and check-in.
6. For a female, must be of non-childbearing potential and therefore must have undergone one of the following sterilization procedures, at least 6 months prior to the first dose:

   1. hysteroscopic sterilization;
   2. bilateral tubal ligation or bilateral salpingectomy;
   3. hysterectomy;
   4. bilateral oophorectomy; or be postmenopausal with amenorrhea for at least 1 year prior to the first dose and follicle-stimulating hormone (FSH) serum levels consistent with postmenopausal status as per PI judgment.
7. A non-vasectomized, male subject must agree to use a condom with spermicide or abstain from sexual intercourse during the study until 90 days beyond the last dose of study drug. (No restrictions are required for a vasectomized male provided his vasectomy has been performed 4 months or more prior to the first dose of study drug. A male who has been vasectomized less than 4 months prior to the first dose must follow the same restrictions as a non-vasectomized male).
8. If male, must agree to not donate sperm from the first dose until 90 days after dosing.
9. Must have the ability to understand and sign a written informed consent form, which must be obtained prior to initiation of study procedures.

Exclusion Criteria:

1. Subject is mentally or legally incapacitated or has significant emotional problems at the time of the screening visit or expected during the conduct of the study.
2. History or presence of clinically significant medical or psychiatric condition or disease in the opinion of the PI.
3. History of any illness that, in the opinion of the PI, might confound the results of the study or poses an additional risk to the subject by their participation in the study.
4. History or presence of alcoholism or drug abuse within the past 2 years prior to the first dose or regular alcohol consumption within 6 months prior to the first dose with an average weekly intake of greater than 21 glasses/units per week for males or 14 glasses/units per week for females, with one unit = 150 mL of wine or 360 mL of beer or 45 mL of 45% alcohol.
5. History or presence of hypersensitivity or idiosyncratic reaction to the study drug(s) or related compounds.
6. History of sensitivity to heparin or heparin-induced thrombocytopenia.
7. Active or latent tuberculosis.
8. Estimated creatinine clearance <80 mL/min at screening.
9. Liver function tests (serum ALT, AST, alkaline phosphatase) and serum bilirubin (total and direct) > ULN.
10. Absolute neutrophil count < 1500 cells/mm3.
11. White blood cell count < 3500 cells/mm3.
12. Haemoglobin levels < 0.5 mg/dL below the lower limit of normal.
13. Seated heart rate is lower than 40 bpm or higher than 99 bpm at screening.
14. Female subjects of childbearing potential.
15. Female subjects who are pregnant or lactating.
16. Positive urine drug or alcohol results at screening or check-in.
17. Positive urine cotinine at screening.
18. Positive results at screening for human immunodeficiency virus (HIV), hepatitis B surface antigen (HBsAg), or hepatitis C antibodies (HCV).
19. Unable to refrain from or anticipates the use of any drug, including prescription and non-prescription medications, herbal remedies, or vitamin supplements beginning approximately 14 days prior to the first dose and throughout the study.. Hormone replacement therapy will not be allowed. After first dosing, acetaminophen (up to 2 g per 24 hours) may be administered at the discretion of the PI or designee.
20. Has been on a diet incompatible with the on-study diet, in the opinion of the PI, within the 28 days prior to the first dose and throughout the study.
21. Donation of blood or significant blood loss within 56 days prior to the first dose.
22. Plasma donation within 7 days prior to the first dose.
23. Exposure to more than four new chemical entities within 12 months prior to first dosing day.
24. The subject has participated in a clinical trial and has received an investigational product within 30 days, or 5 half-lives of the investigational product (whichever is longer) of the first dose of study drug in the current study.
25. Any condition or circumstance, in the opinion of the PI, which may make the subject unlikely to complete the study or comply with study procedures and requirements, or may pose a risk to the subject's safety.
26. Subject has recent history (within 2 weeks of Day -1) of less than 1 bowel movement every 2 days.
27. Subject has recent history (within 2 weeks of Day -1) of abnormal bowel movements, such as diarrhea, loose stools, or constipation.

    Stage 1 Only:
28. Is lactose intolerant.

Ages: 19 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2018-03-20 (Actual); Primary Completion 2018-09-26 (Actual); Study Completion 2018-10-03 (Actual)

PRIMARY OUTCOMES:
The number and severity of treatment emergent adverse events (TEAEs) | 7 days after the last dose
  To assess the safety and tolerability of single and multiple ascending oral doses of BBT-401-1S in healthy adult subjects.

SECONDARY OUTCOMES:
Maximum plasma concentration (Cmax) | 72 hours after the last dose
  To assess Cmax of single and multiple ascending oral doses of BBT-401-1S in healthy adult subjects.
Area under the curve (AUC) | 72 hours after the last dose
  To assess AUC of single and multiple ascending oral doses of BBT-401-1S in healthy adult subjects.
Maximum plasma concentration (Cmax) under fed conditions | 72 hours after the last dose
  To assess Cmax of single oral dose under fed conditions
Area under the curve (AUC) under fed conditions | 72 hours after the last dose
  To assess AUC of single oral dose under fed conditions

CONTACTS AND LOCATIONS:
Locations (1):
- Celerion, Lincoln, Nebraska, United States